CLINICAL TRIAL: NCT04904094
Title: Algorithms for Patient-specific Treatment Planning in Cerebral Palsy Based on the Muscle and Tendon Architecture - Homebased (6-week) Stretching Intervention in Children With Spastic Cerebral Palsy
Brief Title: Homebased (6-week) Stretching Intervention in Children With Spastic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); University Ghent (Other); Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s59945_B
Record Dates: First submitted 2020-12-18; First posted 2021-05-27 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Spastic Cerebral Palsy
Keywords: cerebral palsy; spastic cerebral palsy; stretching intervention; muscle morphology; range of motion; stiffness; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: We will include patients who receive casting at the lower limb for the intervention group. Patient with no indication for treatment will be asked for participation in the control group. The children in the control group will continue their usual care or normal routine treatment, i.e. physiotherapy and orthotic devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This group will receive casting of the lower limb for approximately 2 weeks combined with a passive stretching program of the knee flexors, followed by a homebased stretching exercise program for the plantar flexors and hamstrings for 4 weeks after casting.
  Interventions: Other: Casting of the lower limb and homebased stretching exercise program.
- Control group (No Intervention): This group will continue their usual care or normal routine treatment, i.e. physiotherapy and orthotic devices.

INTERVENTIONS:
Other: Casting of the lower limb and homebased stretching exercise program. — Lower leg casting in combination with removable upper leg casts for approximately 2 weeks and stretching exercises during casting and 4 weeks after casting.
  Arms: Intervention group

SUMMARY:
This study will investigate the effect of a 6-week stretching intervention, consisting of a combination of a 2-week casting period and a home-based stretching program of the plantar flexors and hamstrings, on muscle and tendon lengths, range of motion, stiffness, and functional muscle strength. The study will include patients with spastic cerebral palsy aged between 4 and 11 years old with a Gross Motor Function Classification Score (GMFCS) level between I and III.

DETAILED DESCRIPTION:
This study will investigate the effect of a 6-week stretching intervention on muscle and tendon lengths, range of motion, stiffness, and functional muscle strength. The program consists of a 2-week casting period of the lower legs and a home-based stretching program of the hamstrings, followed by a 4-week stretching program of both the plantar flexors and hamstrings.

The aim is twofold: (1) determine whether a 6-week stretching program for the plantar flexors and knee flexors leads to changes in the morphological muscle and tendon properties of the medial gastrocnemius and semitendinosus, ankle and knee range of motion, muscle strength, gait and gross motor function; and (2) determine the correlation between baseline morphological muscle and tendon properties and the changes in the primary outcome parameters (ankle range of motion and stiffness).

The program will start with a 2-week period of stretching casts for the ankle plantar flexors, combined with a passive stretch program for the hamstrings, followed by a passive and active stretch program for both muscle groups for the remaining 4 weeks. The durations and frequencies for passive and active stretching are based on guidelines published by our own research group and on programs applied by previous research. The program will be set-up as a supervised home-based program on top of the usual care. The morphological muscle and tendon parameters, strength, spasticity, stiffness as well as gross motor function will be assessed before and after the entire 6-week stretching program. At the time of cast removal (after 2 weeks), only the morphological muscle and tendon parameters will be evaluated.

This study includes an intervention and control group which will be group-matched based on diagnosis, GMFCS level and age. The study will include patients with spastic cerebral palsy between 4 and 11 years old and a GMFCS level between I and III. Thirty children with a clinical indication for casting of the lower limb will be included in the intervention group and 30 children without an indication for a specific intervention will be included in the control group. Children in the control group will continue their usual care or normal routine treatment, i.e. physiotherapy and orthotic devices.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of spastic cerebral palsy
* Aged 4-12 years
* GMFCS levels I-III (GMFCS = Gross Motor Function Classification Score, expressing the overall functional level of impairment)
* Sufficient cooperation to comprehend and complete the test procedure
* Indication for casting of the lower limb

Exclusion Criteria:

* Non-ambulatory
* Botulinum toxin A injections six months prior to enrollment
* Lower limb surgery two years prior to enrollment
* Selective dorsal rhizotomy as treatment history
* Presence of ataxia or dystonia
* Cognitive problems that impede measurements
* Severe co-morbidities (severe epilepsy, non-correctable visual impairment, autism spectrum disorders, mental problems that prevent comprehensiveness of the tasks)

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in muscle belly and tendon length of the medial gastrocnemius and semitendinosus | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Estimation of the muscle belly and tendon length by 3D freehand ultrasonography. The primary outcome will be the muscle belly/tendon length ratio.
Change of range of motion of the ankle and knee joint | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Evaluation by an instrumented spasticity assessment
Change of range of motion of the ankle and knee joint | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Evaluation by goniometry

SECONDARY OUTCOMES:
Change in muscle neural (spasticity) and non-neural (stiffness) hyper-resistance | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Evaluation of muscle spasticity and stiffness by an instrumented spasticity assessment
Change in functional muscle strength | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Evaluation of functional muscle strength by the Adapted Functional Strength measure
Change in muscle echointensity | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Estimation of the echointensity by 3D freehand ultrasonography
Change in muscle volume | Between baseline, casting removal (2 to 4 weeks after baseline) and 6 to 8 weeks after baseline.
  Estimation of muscle volume by 3D freehand ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, prof. dr., Study Director — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franki I, Desloovere K, De Cat J, Feys H, Molenaers G, Calders P, Vanderstraeten G, Himpens E, Van Broeck C. The evidence-base for basic physical therapy techniques targeting lower limb function in children with cerebral palsy: a systematic review using the International Classification of Functioning, Disability and Health as a conceptual framework. J Rehabil Med. 2012 May;44(5):385-95. doi: 10.2340/16501977-0983. PMID 22549646
- [Background] Lee GP, Ng GY. Effects of stretching and heat treatment on hamstring extensibility in children with severe mental retardation and hypertonia. Clin Rehabil. 2008 Sep;22(9):771-9. doi: 10.1177/0269215508090067. PMID 18728130
- [Background] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387
- [Background] Pin T, Dyke P, Chan M. The effectiveness of passive stretching in children with cerebral palsy. Dev Med Child Neurol. 2006 Oct;48(10):855-62. doi: 10.1017/S0012162206001836. PMID 16978468
- [Background] Theis N, Korff T, Kairon H, Mohagheghi AA. Does acute passive stretching increase muscle length in children with cerebral palsy? Clin Biomech (Bristol). 2013 Nov-Dec;28(9-10):1061-7. doi: 10.1016/j.clinbiomech.2013.10.001. Epub 2013 Oct 10. PMID 24210836
- [Background] van den Noort JC, Bar-On L, Aertbelien E, Bonikowski M, Braendvik SM, Brostrom EW, Buizer AI, Burridge JH, van Campenhout A, Dan B, Fleuren JF, Grunt S, Heinen F, Horemans HL, Jansen C, Kranzl A, Krautwurst BK, van der Krogt M, Lerma Lara S, Lidbeck CM, Lin JP, Martinez I, Meskers C, Metaxiotis D, Molenaers G, Patikas DA, Remy-Neris O, Roeleveld K, Shortland AP, Sikkens J, Sloot L, Vermeulen RJ, Wimmer C, Schroder AS, Schless S, Becher JG, Desloovere K, Harlaar J. European consensus on the concepts and measurement of the pathophysiological neuromuscular responses to passive muscle stretch. Eur J Neurol. 2017 Jul;24(7):981-e38. doi: 10.1111/ene.13322. Epub 2017 May 29. PMID 28557247